CLINICAL TRIAL: NCT01790399
Title: IDENTIFICATION OF SENTINEL NODE(S) BY SENTIMAG® /SIENNA+ IN BREAST CANCER: FEASIBILITY STUDY
Brief Title: IDENTIFICATION OF SENTINEL NODE(S) IN BREAST CANCER
Acronym: SENTIMAG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Sysmex America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SENTIMAG-1213
Record Dates: First submitted 2013-02-08; First posted 2013-02-13 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2013-08

CONDITIONS: BREAST CANCER
Keywords: SENTINEL NODE
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Identification of sentinel node(s) (Experimental)
  Interventions: Procedure: Excision of sentinel node(s)

INTERVENTIONS:
Procedure: Excision of sentinel node(s) — Excision of sentinel node(s) using SENTIMAG / SIENNA + in addition to the usual method (blue and /or radioactive product)

SUMMARY:
The study is based on the identification of sentinel node(s) by SENTIMAG / SIENNA + in addition to the usual method (blue and /or radioactive product). This is a feasibility study

DETAILED DESCRIPTION:
* Identification of Sentinel node(s)

  1. Step 1: Identification using the technique Nanocis Sub-areolar injection of Tc99m-Nanocis ® the day before or the day of surgery
  2. Step 2: Identification using the technique SentiMag ® / Sienna+ Injection Sienna + ™ should be done just after induction of anesthesia and before the injection of Patent Blue dye
  3. Step 3: Identification using the technique of Patent Blue Dye or Lymphotropic dye injection or Patent Blue is performed after induction of anesthesia, the injection and production Sienna + ™, the operating theater by the surgeon
* Detection of Sentinel node(s)

  1. Step 1: probe SentiMag ® (study)
  2. Step 2: hand probe gamma radiation detection and / or colorimetric detection (standard)
* Sentinel node's excision of radioactive and / or blue and / or magnetic (colored brown-brown)
* After the procedure:

Characterization of the size and weight of lymph nodes, histological and / or molecular OSNA and linking nodal status with the detection rate of sentinel nodes for each technique.

NB: In case of synchronous bilateral cancer, 2 records are possible

ELIGIBILITY:
Inclusion Criteria:

* Patient with invasive breast cancer or microinfiltrant proven by cytology and histo-or whatever the histological type
* cT0/cT1/cT2 (up to 5 cm) CN0 clinical and / or ultrasound and without prior treatment (chemotherapy or neoadjuvant hormone )
* Age greater than or equal to 18
* Reporting of breast surgery and axillary staging of sentinel lymph node
* Using effective contraception (BHCG negative)
* Patient affiliated with a health insurance
* Consent signed by the patient

Exclusion Criteria:

* T3 or T4 tumors (> 5 cm, cutaneous or muscle inflammation or cancer)
* Presence of a clinically suspicious axillary adenopathy or imaging
* Tumors bifocal or multifocal known before Surgery
* History of breast surgery or axillary
* Patient metastatic
* Patient with a cons-indication anesthesia and / or surgery
* Intolerance or hypersensitivity to the compounds or iron dextran or superparamagnetic iron oxide or to Patent blue dye in centers where it is commonly used
* Patient can not receive a radioactive isotope to the sentinel lymph node resection
* Allergy radioactive product
* Chronic iron overload
* Pacemaker or other implantable device in the chest wall
* Failure to submit to medical study for geographical, social or psychological
* Patient deprived of liberty or under guardianship
* Pregnant or lactating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Sentinel node(s)detected with new technical | The day of surgery
  Idenfication 's rate of sentinel nodes detected with new technical(SentiMag ® / Sienna + TM)

SECONDARY OUTCOMES:
Detected node(s) for each method(standard and new) | The day of surgery
  Proportion of detected nodes for each method(standard and new)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis MD HOUPEAU, Study Director — Centre Oscar Lambret
Locations (4):
- France (4):
  - Centre Oscar Lambret, Lille
  - Centre Eugène Marquis, Rennes
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy